CLINICAL TRIAL: NCT04482556
Title: Comparison of the Q-NRG+ Indirect Calorimetry Device Versus the V(Max) Encore Device in Mechanically Ventilated Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Ben D. Albert, MD, Director, Critical Care Medicine Fellowship Program, Boston Children's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-P00033440
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Calorimetry, Indirect; Oxygen Consumption; Metabolism; Mechanical Ventilation
Keywords: Pediatrics; Indirect Calorimetry; Enteral Nutrition; Metabolism; Critical Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Q-NRG+ Indirect Calorimetry Device (Other): Q-NRG+ device will be compared to current V(max) device in each enrolled patient in subsequent, alternating fashion.
  Interventions: Device: Q-NRG+ Indirect Calorimetry Device
- V(max) Encore Indirect Calorimetry Device (Other): V(max) Encore device, currently institution's standard device, will be compared to Q-NRG+ device in each enrolled patient in subsequent, alternating fashion.
  Interventions: Device: V(max) Encore Indirect Calorimetry Device

INTERVENTIONS:
Device: Q-NRG+ Indirect Calorimetry Device — The two indirect calorimetry devices will be tested in an alternating fashion for each enrolled patient. Each enrolled patient subsequently will alternate in which device is tested first.
  Arms: Q-NRG+ Indirect Calorimetry Device
Device: V(max) Encore Indirect Calorimetry Device — The two indirect calorimetry devices will be tested in an alternating fashion for each enrolled patient. Each enrolled patient subsequently will alternate in which device is tested first.
  Arms: V(max) Encore Indirect Calorimetry Device

SUMMARY:
The overarching aim of this proposal is to examine the feasibility of the Q-NRG+ indirect calorimetry device and its agreement with (Vmax) Encore indirect calorimetry device in mechanically ventilated children. The overall hypothesis of this study is that the Q-NRG+ will provide minute-to-minute oxygen consumption (VO2) and carbon dioxide production (CO2) measurements that are in agreement with those obtained by the standard indirect calorimetry device currently used at our institution (Vmax Encore).

DETAILED DESCRIPTION:
Indirect calorimetry allows accurate measurement of energy expenditure in this population but current technology is cumbersome and time-consuming, and has many limitations that exclude a majority of criticaly ill children. A new device was recently developed to address some of the limitations of IC devices and is widely endorsed for IC measurements in critically ill adults. The Q-NRG+ IC device incorporates an easier gas calibration technique to facilitate faster start up, and a micro-mixing chamber (2ml) allows rapid achievement of steady state gas exchange measurement. The device may address some of the current barriers for the use of indirect calorimetry in critically ill children. A device with short calibration time and reliable measurements could enhance the ability of clinicians to deliver individualized energy prescriptions for patients.

Description of Study Treatments

Following informed consent, the following steps will be followed for the study procedure:

1. The two testing indirect calorimetry devices will be tested in an alternating fashion for each enrolled patient, therefore it will be decided the V(max) will be tested first in the first enrolled patient then the Q-NRG+ second. Each enrolled patient subsequently will alternate in which device is tested first.
2. The first device will be connected to the patient, after calibration, and data collection will begin for a maximum duration of 30 minutes.
3. At the end of the first testing period, the first device will be disconnected and the second device will be connected to the study patient.
4. Data collection for the second device will then begin for a maximum duration of 30 minutes.
5. At the end of the testing period, the data collected for the V(max) device will be discussed with the parents and the clinical team. Data collected from the Q-NRG+ will not be shared with the clinical team or family as this device is still being investigated in the pediatric population.
6. The study will then conclude.

Definitions of Outcomes/Endpoints The primary variables to be collected are steady state measurements of VO2 and VCO2 from both indirect calorimetry devices. Steady state will be defined as a period of greater than five minutes with coefficient of variation of the VO2 and VCO2 measurements of less than 10%. If steady state is not achieved, energy calculations will not be included in data analysis. Secondary variables to be collected include total time to obtain indirect calorimetry measurement, from arrival at the bedside to completion of the study. Steady state conditions will be defined using existing institutional practice.

Data Collection Methods and Assessments Descriptive characteristics will also be collected for each patient including age, weight, height, diagnosis, severity of illness, length of ICU stay, vital signs, and ventilator settings. We will also collect endotracheal tube size, presence of cuff, leak percentage. We will also collect information about medications, including inotropes and vasopressors, sedation medications (as well as SBS score) and nutrition parameters. Markers of inflammation, WBC and CRP will be collected from the patient chart.

Statistical Analysis Descriptive statistics will be computed for measured REE, VO2 and VCO2 and Bland-Altman analysis will be utilized to quantify the mean bias and limits of agreement between devices. Acceptable limits of agreement between the devices will be +/- 20%. VO2, CO2 will be reported as means (SD). The time to steady state and total time of IC measurement will be compared using a T-test (if normally distributed) or Mann-Whitney U-test (if not normally distributed).

ELIGIBILITY:
Inclusion Criteria:

* Children mechanically ventilated with endotracheal tube of tracheostomy in standard ventilatory modes such as SIMV-PC, SIMV-VC or PRVC
* Age > 10 years AND weight > 10kg
* FIO2 < 60%
* PEEP < 8
* ETT leak < 10%
* The attending physician of record plans to order indirect calorimetry and considers research activity safe

Exclusion Criteria:

* Hemodynamic instability (hypotension according to PALS/ACLS formula or requiring 2 or greater vasoactive infusions)
* Presence of chest tubes with ongoing air leak
* Patients requiring ECMO support
* Patients undergoing end-of-life care
* Primary provider declines enrollment.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean bias and limits of agreement between measured oxygen consumption (VO2) and carbon dioxide elimination (VCO2) in mechanically ventilated children assessed using the Q-NRG+ indirect calorimetry device and the V(max) Encore indirect calorimetry device. | 1 hour/participant
  In mechanically ventilated children, we will describe the mean bias and limits of agreement in measurements using both indirect calorimeters. Our hypothesis is that the measurement of oxygen consumption (VO2) and carbon dioxide production (VCO2) with the 2 devices will have a low mean bias and will be within clinically acceptable limits of agreement.
Calculated total testing time, including calibration, required to complete a steady state indirect calorimetry measurement using the Q-NRG+ device and the V(max) Encore. | 1 hour/participant
  Total time lapsed, including time for patient data input, warm-up, calibration, and gas exchange measurements in steady state will be recorded. Our hypothesis is that the time required to obtain energy expenditure with Q-NRG+ device will be significantly shorter as compared to the Vmax Encore device.

CONTACTS AND LOCATIONS:
Overall Officials: Nilesh M Mehta, MD, Study Director — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No